CLINICAL TRIAL: NCT05621577
Title: Socio-Demographic - Dental & Respiratory Changes of Obstructive Sleep Apnea (OSA) Patients Treated With Mandibular Advancement Device (MAD) of Samples in Erbil City
Brief Title: Obstructive Sleep Apnea Patients Treated With Mandibular Advancement Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Haval Jalal Rasheed, assistant lecturer, Hawler Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sleep apnea orthodontics
Record Dates: First submitted 2022-11-07; First posted 2022-11-18 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Sleep Apnea, Obstructive
Keywords: orthodontic
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Occlusal Splints

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mandibular advancing device (Other): using mandibular advancement device for treatment of obstructive sleep apnea
  Interventions: Device: MANDIBULAR ADVANCEMENT DEVICE

INTERVENTIONS:
Device: MANDIBULAR ADVANCEMENT DEVICE — orthodontically treating obstructive sleep apnea

SUMMARY:
The purpose of this study is to evaluate efficacy of mandibular advancement device (MAD). on treating obstructive sleep apneas, symptoms, Apnea/Hypopnea Index (QHI) and the Respiratory Arousal Index (AHI/REI) and peripheral capillary oxygen saturation (SpO2) Range, PULSE in patients with mild to moderate obstructive sleep apnea/hypopnea syndrome, and evaluating potential dental side effects

DETAILED DESCRIPTION:
The primary oral appliance (OA) used in obstructive sleep apnea (OSA) treatment is the mandibular advancement device (MAD). MADs may be either an over-the-counter stock device or customized for individual patients. MADs come in various designs and materials, but most comprise upper and lower splints mounted over the dentition as either a 1-piece monoblock or a 2-piece biblock Connectors or blocks relate the upper and lower splints in a biblock to protrude the mandible in a forward position during sleep.

Although the efficacy of oral appliances has been proved, the relationship to the nature of airway enlargement in patients with OSA has not yet been clearly demonstrated.

The aim of this study is therefore to evaluate the efficacy mandibular repositioning appliance reduces sleep apneas symptoms with mild to moderate obstructive sleep apnea . Secondary outcomes include the dental side effects of such appliance. At baseline and after 4 month's treatment, This study will be conducted to estimate frequency of OSA on population sample from Erbil study, in addition trying to evaluate the efficiency of MAD on some patients who are diagnosed with OSA.

ELIGIBILITY:
Inclusion Criteria:

1. sample will be taken from Kurdish population in Erbil city.
2. Obstructive sleep apnea, apnea-hypopnea index of <30 with excessive daytime sleepiness

Exclusion Criteria:

1. People with problems in nasal part of airway.
2. People with cleft lip and palate
3. Patient who did tonsillectomy and / or other pharyngeal operations.
4. People who take any kind of sleep medication.
5. Temporomandibular Disorders.
6. People with periodontal disease.
7. Less than 8 teeth/ arch.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-05 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
measuring polysomnography record changes pre and post using appliance | 6 months
  comparing polysomnography readings before and after using MAD to evaluate appliance efficacy

SECONDARY OUTCOMES:
dental side effects | 6 months
  digital dental models before and after treatment to evaluate side effects

CONTACTS AND LOCATIONS:
Overall Officials: Zana Omer, Assist.Prof, Study Director — Hawler Medical University
Locations (1):
- Hawler medical university, Erbil, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Randerath W, Verbraecken J, de Raaff CAL, Hedner J, Herkenrath S, Hohenhorst W, Jakob T, Marrone O, Marklund M, McNicholas WT, Morgan RL, Pepin JL, Schiza S, Skoetz N, Smyth D, Steier J, Tonia T, Trzepizur W, van Mechelen PH, Wijkstra P. European Respiratory Society guideline on non-CPAP therapies for obstructive sleep apnoea. Eur Respir Rev. 2021 Nov 30;30(162):210200. doi: 10.1183/16000617.0200-2021. Print 2021 Dec 31. PMID 34853097
- [Background] Keim RG, Graham JW, Palomo JM, Shoaf SC, Tanguay D. Obstructive sleep apnea treatment in orthodontic practices. J Clin Orthod. 2022 Jan;56(1):23-33. No abstract available. PMID 35704888
- [Background] Keim RG. The orthodontist and obstructive sleep apnea. J Clin Orthod. 2022 Jan;56(1):8. No abstract available. PMID 35704890
- [Background] Gambino F, Zammuto MM, Virzi A, Conti G, Bonsignore MR. Treatment options in obstructive sleep apnea. Intern Emerg Med. 2022 Jun;17(4):971-978. doi: 10.1007/s11739-022-02983-1. Epub 2022 Apr 23. PMID 35460431
- [Background] Damian A, Gozal D. Innovations in the Treatment of Pediatric Obstructive Sleep Apnea. Adv Exp Med Biol. 2022;1384:339-350. doi: 10.1007/978-3-031-06413-5_20. PMID 36217094
- [Background] Ho ACH, Savoldi F, Wong RWK, Fung SC, Li SKY, Yang Y, Gu M. Prevalence and Risk Factors for Obstructive Sleep Apnea Syndrome Among Children and Adolescents with Cleft lip and Palate: A Survey Study in Hong Kong. Cleft Palate Craniofac J. 2023 Apr;60(4):421-429. doi: 10.1177/10556656211068306. Epub 2021 Dec 23. PMID 34939456
- [Background] Triggs A, Roberson G, Chaudhry K, Subramani K. Screening for obstructive sleep apnea by orthodontists in the United States - A survey study. J Clin Exp Dent. 2022 Aug 1;14(8):e625-e632. doi: 10.4317/jced.59708. eCollection 2022 Aug. PMID 36046169
- [Background] Bozzini MF, Di Francesco RC, Soster LA. Clinical and anatomical characteristics associated with obstructive sleep apnea severity in children. Clinics (Sao Paulo). 2022 Nov 1;77:100131. doi: 10.1016/j.clinsp.2022.100131. eCollection 2022. PMID 36334493
- [Result] Bariani RCB, Bigliazzi R, Cappellette Junior M, Moreira G, Fujita RR. Effectiveness of functional orthodontic appliances in obstructive sleep apnea treatment in children: literature review. Braz J Otorhinolaryngol. 2022 Mar-Apr;88(2):263-278. doi: 10.1016/j.bjorl.2021.02.010. Epub 2021 Mar 14. PMID 33757756